CLINICAL TRIAL: NCT01351532
Title: Behavior Change on Oral Cancer Patients After a Localized Behavior Change Model Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMR100-IRB-063
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Lifestyle counseling, smoking cessation drug (Experimental)
  Interventions: Behavioral: smoking cessation program
- Lifestyle counseling (Active Comparator)
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: smoking cessation program — cross-theoretical model integrating smoking cessation counseling, smoking cessation drug utilization, physician interview and telephone counseling persuasion,
  Arms: Lifestyle counseling, smoking cessation drug
Behavioral: Lifestyle counseling — ross-theoretical model integrating smoking cessation counseling,physician interview and telephone counseling persuasion
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this research is to apply this smoking cessation program on oral cancer patients, and to analyze the effectiveness of it.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of oral cancer
* current smoker

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taichung, Taiwan